CLINICAL TRIAL: NCT06811077
Title: As Part of Therapeutic Education for Patients Registered At the Chronic Pain Consultation
Brief Title: Evaluation of Individual Health Coaching Sessions Provided by a Patient Expert As Part of Therapeutic Education for Patients Registered At the Chronic Pain Consultation
Acronym: COADOL
Status: Recruiting | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: COADOL
Record Dates: First submitted 2025-01-30; First posted 2025-02-06 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- individual coaching
  Interventions: Other: individual coaching

INTERVENTIONS:
Other: individual coaching — in addition to group therapeutic education, the patient participates to individual coaching session and answers several Patient Reported Outcome to assess his wellbeing

SUMMARY:
Chronic pain is defined as a persistent sensory and emotional experience, lasting for more than three months, and often resistant to treatment. It can result from various conditions, including life-threatening diseases, accidents, or therapeutic procedures like surgery or chemotherapy. Chronic pain significantly impacts a patient's physical and psychological well-being, often leading to body image issues and functional deterioration in daily activities, both at home and at work or school. The World Health Organization recognized chronic pain as a disease in 2019. Chronic pain patients must adapt to their condition, acquiring new skills and knowledge through therapeutic education. Group sessions, a key part of therapeutic education, help break the isolation felt by many patients, fostering shared experiences and mutual support. Since 2015, the Saint-Joseph Hospital's chronic pain consultation has offered group education workshops, inspired by those at the Pitié-Salpêtrière hospital in Paris. However, many patients struggle to apply new skills independently after these workshops. In response, individualized coaching was introduced in 2020. This approach, led by a health coach who is also an expert patient, provides personalized support to help patients set and achieve realistic goals, fostering active engagement in their lives through tailored strategies and ongoing support.

The main aim of this pilot study is to assess the quantitative and qualitative contribution of personalized support by an "expert patient" chronic pain coach (individual coaching), on the functional and emotional impact and emotional impact of their pain, in patients followed up in a chronic pain consultation and having group therapeutic education workshops.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years
* Patients followed in chronic pain consultations referred to the therapeutic education workshops
* Patient affiliated with a health insurance plan
* French-speaking patient
* Patient capable of giving oral, informed, and explicit consent

Exclusion Criteria:

* Patient with psychiatric disorders making inclusion in group workshops impossible
* Patient unwilling to participate in individual coaching sessions Patient under guardianship or curatorship Patient deprived of liberty Patient under legal protection Pregnant or breastfeeding patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed in chronic pain consultations referred to the therapeutic education workshops
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
BPI (Brief Pain Inventotry ) | enrollment, 4, 6 and 12 months
  evaluation of functional and emotional impact of pain assess with the Brief Pain inventory on a scale from 0 to 10

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Saint Joseph, Paris, France, France

IPD SHARING:
Plan to Share IPD: No